CLINICAL TRIAL: NCT05133947
Title: A Clinical Study Examining Intraepidermal Nerve Fiber Density (IENFD) in Patients With Chemotherapy-induced Peripheral Neuropathy (CIPN) Compared With Healthy Subjects
Brief Title: Pre-study to Evaluate IENFD Induction in Patients With Taxane-induced CIPN
Status: Completed | Type: Observational
Sponsor: Beijing 3E-Regenacy Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: BCRG-CN-001
Record Dates: First submitted 2021-11-04; First posted 2021-11-24 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2021-11

CONDITIONS: Peripheral Nervous System Diseases
MeSH Terms: conditions — Peripheral Nervous System Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CIPN patient: Patient with CIPN symptom
  Interventions: Other: Non interventional
- Healthy subject: Healthy subject
  Interventions: Other: Non interventional

INTERVENTIONS:
Other: Non interventional — Non interventional

SUMMARY:
This is a non-interventional study examining IENFD levels in patients with CIPN after taxane chemotherapy and in age-matched healthy subjects.

DETAILED DESCRIPTION:
This is a non-interventional study examining IENFD levels in patients with CIPN after taxane chemotherapy and in age-matched healthy subjects. After the subjects sign the informed consent, the study physicians will judge the inclusion and exclusion criteria. Subjects meeting the inclusion requirements will register at the study center according to the requirements of the study physicians, and skin samples will be collected by specialized researchers.

ELIGIBILITY:
Inclusion Criteria:

Received taxane adjuvant chemotherapy for breast cancer for curative purposes and completed chemotherapy before entering the study; Persistent peripheral neuropathy of the lower extremities;

CIPN Severity:

The presence of at least one of the following symptoms on both lower extremities in a gloved and sock glove pattern: pain or burning, numbness, or tingling.

Examination of the lower extremities showed needling loss of both legs; Neurological symptoms occur after exposure to taxane and cannot be attributed to any other neurological disease; NRS rating ≥ 4.

Exclusion Criteria:

Pregnant or lactating women. Presence of any neuropathy other than CIPN. According to the investigator's judgment, there are skin diseases in the affected skin area that may interfere with the evaluation of neuropathic pain symptoms, or diseases at the skin biopsy site that may affect the epidermal nerve morphology, or other factors.

The presence of non-CIPN pain may interfere with study evaluation and/or peripheral neuropathic pain self-assessment.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 18-70 years old CIPN Patients and healthy subjects.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
IENFD | 2021.10~2022.6
  IENFD change between CIPN patients and healthy subjects

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojiao Li, Principal Investigator — China
Locations (1):
- Bethune First Hospital Of Jilin University, Jilin, China

IPD SHARING:
Plan to Share IPD: No